CLINICAL TRIAL: NCT00745524
Title: Screening for Attention-deficit/Hyperactivity Disorder (ADHD) in Adolescent and Adult High Risk Populations
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200801026R
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention-deficit hyperactivity disorder; adolescent; adult; high risk population; functional impairment; quality of life
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to investigate the prevalence of ADHD and other psychopathology, and current function and life quality among several high risk populations of imprisoned adults and adolescents who receive special resources in school or dropout from school.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is a common (5-10%) childhood-onset neuropsychiatric disorder worldwide among children and adolescents with 50- 60% persistence to adulthood (3-4%). Individuals with ADHD have been reported to have higher risk of school failure, conduct problems, antisocial behaviors, legal problems, substance use problems and other psychiatric comorbidities, and face many difficulties of the interpersonal relationship, occupation and family in every day life. Despite plenty of researches reported in the west countries, we have limited information in Taiwan about adult ADHD and the associated impact on the function and quality of life of the affected individuals. For the perspective of public health, it's mandatory to collect information from the high risk populations of ADHD for further policy establishment to prevent further impact on individuals, families, and society in Taiwan.

This study target on two populations: (1) imprisoned adults (2) adolescents with problems in school and followed by three private charitable organizations. Each population is assessed by the instruments for ADHD symptoms (ASRS and SNAP-IV), psychopathology (ASRI and/or YSR and CBCL), and academic/social/occupational /family function (WFIRS-S, WFIRS-P). Adult population is also checked for the quality of life (AAQoL). We will recruit the community-based controls matching with sex and age is assessed with the same instruments.

We anticipate that this study will provide the primitive data on the prevalence of ADHD and other psychopathology, academic/occupational/social/family function, quality of life of adolescent and adult patients in the high risk populations, will evaluate the difference between adults in prison, adolescents dropping out from school, and their community controls with regards to symptomatology, quality of life, and function; and young psychiatric researchers will learn to collect data, conduct statistical analysis, and prepare the manuscript. Our findings should have clinical implication in assessing adults and adolescents at high risk of ADHD and provide the reference data for future public health policy planning regarding early identification of ADHD at childhood and intervention program to offset the adverse social and academic/occupational sequalae of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* The adult subjects aged 20~65 form National Tainan Prison are recruited.
* The adolescent subjects aged 13~19, drop out from school or receiving special services, followed by three private charitable organizations are recruited.
* The controls will be recruited according to the structure of sex and age of the cases.

Exclusion Criteria:

* In the major depressive episode, comorbid with severe anxiety disorders or during substance intoxication or withdrawal, or during the acute psychotic episode at the time of evaluation.
* With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Imprisoned adults; adolescents with problems in school and followed by three private charitable organizations; community sample
Sampling Method: Non-Probability Sample
Enrollment: 1910 (Actual)
Dates: Start 2008-02; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Tainan Prison, Tainan
  - Tainan Family Educational Center, Tainan